CLINICAL TRIAL: NCT02556073
Title: The Use of ﬂuticasone Propionate/Salmeterol Inhaler With Integrated Dose Counter and Smartphone Self Management to Improve Airway Inflammation and Asthma Control
Brief Title: ICS/LABA Combination With Integrated Dose Counter and Smartphone APP to Improve Asthma Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140218
Record Dates: First submitted 2014-11-25; First posted 2015-09-22 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Asthma
Keywords: asthma control; adherence; asthma self management plan; airway inflammation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): "Usual care" means that intervention by fluticasone/salmeterol 125/25 2 puffs bid plus salbutamol as needed acts as asthma controller and patients will be scheduled to revisit clinics.
  Interventions: Drug: usual care
- Usual care+Smartphone action (Experimental): Intervention by fluticasone/salmeterol 125/25 2 puffs bid plus salbutamol as needed and Smartphone action, which provides the real-time health information of surroudings and actively remind the patients to use controller.
  Interventions: Other: Smartphone action; Drug: usual care

INTERVENTIONS:
Other: Smartphone action — Smartphone applications (Apps) can provides a platform not only to share health information at the point-of-living, including health assessments, personalized health plans, but also to remind the patients' medication adherence regularly. With the application of modern smartphone-based asthma self management deserves further investigation to improve asthma control.
  Other Names: asthma controller+Smartphone self-management
  Arms: Usual care+Smartphone action
Drug: usual care — fluticasone/salmeterol 125/25 ug/puff, 2 puff bid plus salmeterol as-needed
  Other Names: asthma controller

SUMMARY:
Poor adherence to asthma controller medication may link to poor asthma outcome. A metered dose device with built-in dose counter helps physicians to monitor drug compliance in asthma patients. Mobile-phone based self management opens a window for better asthma control. The present study aims to investigate the relationship between the adherence to controller medication of combined inhaled corticosteroid/long acting beta2-agonists, assessing by integrated dose counter, and the level of airway inflammation and asthma control. Moreover, the investigators also use a new asthma self-management Apps to enhance drug compliance. With the application of the new, easily available tools, the investigator expect to increase adherence rates, and hence, to reduce airway inflammation and improve the level of asthma control.

DETAILED DESCRIPTION:
The study will be conducted as a prospective, observational, open labeled, randomized trial in a single center (Taipei Veterans General Hospital). After screening, the enrolled patients will be randomized to either routine care or Smartphone self management group. In the routine care group, the patient will be treated as routine practice as a real-world setting. No additional intervention will be done. In the Smartphone self management group, an asthma self management Apps (My asthma App, GlaxoSmithKline, Chinese version, or Line), which provides multiple function, including health information (real-time weather condition, air pollution index) at the point-of-living, personalized health assessments (asthma control test, peak flow rate) and interactive action plans (green, yellow, and red light), and regular reminding for controller administration, will be downloaded to the participant's Smartphone. The participant will be educated to operate the Apps to improve asthma control. Participants in both groups will use identical controller (Sal/flu 2 inhalations twice daily plus as-needed rescue ventolin) and will be scheduled to follow up for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic asthmatics free of controller medication for at least 3 months
2. Aged from 20 to 70 years
3. Life-long smoking index < 10 pack-years

Exclusion Criteria:

1. COPD, clinically overt bronchiectasis, lung cancer, active tuberculosis, or other known specific pulmonary disease.
2. A chest X-ray indicating diagnosis other than asthma that might interfere with the study.
3. Major disease abnormalities are uncontrolled on therapy.
4. Alcohol or medication abuse.
5. Patients had lower respiratory tract infections or received systemic steroid in the 4 weeks prior to the commencement of study.
6. Unable or unwilling to comply with all protocol
7. Unable to use Smartphone

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Changes of airway inflammation profile | Changes of airway inflammation profile from baseline at 24 weeks
  measurement including exhaled NO, cell counts and mediator in induced sputum before (baseline, wk0) and after treatment (wk 24)

SECONDARY OUTCOMES:
changes of scores of asthma control questionnaire | Changes of scores of asthma control questionnaire from baseline at 24 weeks
  scores of questionnaire of asthma control test (ACT)
Changes of lung function parameters | Changes of lung function parameters (FEV1, FVC) from baseline at 24 weeks
Numbers of rescue medication use | Total numbers of rescue medication use during 24-week period

CONTACTS AND LOCATIONS:
Overall Officials: Kang-Cheng Su Su, Md. MS, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan